CLINICAL TRIAL: NCT00002780
Title: INFUSION OF ACTIVATED T CELLS AND LOW DOSE INTERLEUKIN 2 COMBINED WITH PERIPHERAL BLOOD STEM CELL TRANSPLANTATION FOR THE TREATMENT OF WOMEN WITH METASTATIC BREAST CANCER: PHASE I/II
Brief Title: Biological Therapy in Treating Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Luke's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064792; STLMC-BRM-9503; NCI-V96-0902
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — aldesleukin; sargramostim; Carboplatin; Cyclophosphamide; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: cytokine therapy
Biological: sargramostim
Drug: carboplatin
Drug: cyclophosphamide
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining different types of biological therapies may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of T cells and interleukin-2 combined with peripheral stem cell transplantation or bone marrow transplantation in treating women who have stage IIIB or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the toxicities of the combination of low dose interleukin-2 (IL-2) sargramostim (GM-CSF), and multiple doses of activated T cells (ATC) following peripheral blood stem cell transplantation in women with stage IIIB or metastatic adenocarcinoma of the breast. II. Evaluate the efficacy of this regimen in these patients.

OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously daily for 5 days prior to peripheral blood stem cell (PBSC) collection or for 2 days prior to bone marrow harvest. Following PBSC collection or bone marrow harvest, patients receive high dose chemotherapy consisting of cyclophosphamide IV, carboplatin IV, and thiotepa IV over days -6 through -3. Patients undergo PBSC transplantation on day 0. Following PBSC transplantation, patients receive multiple doses of monoclonal antibody OKT3 activated T lymphocytes IV over 1 hour between days 1 and 65, continuous low dose interleukin-2 (IL-2) IV over days 1-65, and sargramostim (GM-CSF) subcutaneously on days 5-21. Patients are followed at day 100, as clinically indicated, and then annually.

PROJECTED ACCRUAL: Approximately 40-60 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented metastatic adenocarcinoma of the breast Concurrent intraductal or lobular carcinoma in situ allowed Bilateral disease allowed Measurable or evaluable recurrent metastatic disease (Stage IIIB or IV) documented by radiograph, CT scan, nuclear medicine scan, or physical exam Tumor must be clinically chemosensitive as documented by a reduction in tumor burden No clinical evidence of brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 50,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin less than 1.5 times normal Hepatitis B surface antigen negative Renal: Creatinine less than 1.8 mg/dL Creatinine clearance normal Blood urea nitrogen (BUN) less than 1.5 times normal Cardiovascular: Ejection fraction at least 45% by MUGA No uncontrolled or significant cardiovascular disease including myocardial infarction (less than 1 year) or congestive heart failure Pulmonary: PFT-FEV1 at least 60% of predicted DLCO and FVC at least 60% of predicted Other: Not pregnant Negative pregnancy test HIV negative No serious medical or psychiatric illness No prior or concurrent malignancy, other than curatively treated carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY: See Disease Characteristics No concurrent hormonal therapy for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1996-05

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- St. Luke's Medical Center, Milwaukee, Wisconsin, United States